CLINICAL TRIAL: NCT04524312
Title: Does Dynamic Congruence Design Improve Gait After Total Knee Replacement in Comparison to Posterior-stabilized One? - Prospective Randomized Controlled Trial
Brief Title: Dynamic Congruence Total Knee Replacement vs Posterior-stabilized
Acronym: K-Mod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, MD, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WarsawMU/kmod
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Osteo Arthritis Knee; Surgery; Joint Diseases
Keywords: osteoarthritis; knee; congruence; posterior-stabilized; cruciate-retaining
MeSH Terms: conditions — Joint Diseases; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee; Biomechanical Phenomena

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will not be informed which type of prosthesis was used in their particular case.
  Outcomes Assessor will not be informed which type of prosthesis was used in particular patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NexGen (Active Comparator): Patients undergoing total knee replacement for treatment of primary knee ostearthritis with use of Zimmer Biomet NexGen prosthesis
  Interventions: Procedure: Total knee replacement; Diagnostic Test: Biomechanics; Device: NexGen Ps or Bioimplanti K-MOD implant
- K-Mod (Active Comparator): Patients undergoing total knee replacement for treatment of primary knee ostearthritis with use of Bioimplanti K-MOD prosthesis
  Interventions: Procedure: Total knee replacement; Diagnostic Test: Biomechanics; Device: NexGen Ps or Bioimplanti K-MOD implant

INTERVENTIONS:
Procedure: Total knee replacement — Participant will undergo total knee replacement performed via anterior parapatellar approach with either Posterior-stabilized or retaining cruciate-retaining with dynamic congruence implant
Diagnostic Test: Biomechanics — Participants will be asked to perform biomechanical assesment before and following surgery at baseline, 6-8 weeks and 6-months postoperatively
Device: NexGen Ps or Bioimplanti K-MOD implant — Participant are randomly allocated to receive one of the NexGen PS or Biomplanti K-MOD total knee implant for treatment of end-stage knee osteoarthritis.

SUMMARY:
This study compares and evaluates differences in movement analysis, patient-reported outcome between patients undergoing total knee arthroplasty with use of either Zimmer Biomet NexGen with posterior stabilization and Bioimplanti K-Mod cruciate-retaining with dynamic congruence

DETAILED DESCRIPTION:
The aim of this study is to assess and compare kinematic and time-space gait parameters in patients after total knee arthroplasty, who will undergo the surgery with the use of either posterior-stabilized (PS) or dynamic congruence (DC) implants.

Materials and methods To this study 56 consecutive patients undergoing total knee arthroplasty will be recruited. Study protocol is designed as a prospective, blinded, parallel-group, superiority trial, with balanced randomization [1:1]. All participants will be operated in single clinical orthopedic department, by single high-volume surgeon, who performed more than 3000 total knee arthroplasties in his professional career.

Before the surgery patients will fulfill the author's questionnaire concerning their age, height and body mass, level of activity and VAS (Visual Analogue Scale).

After the surgery 1 to 3 years postoperatively three-dimensional gait analysis will performed with use of BTS SMART device. This device uses passive markers technology and registers the movement by six cameras. To perform full gait analysis several data concerning patients anthropometry will be collected (lower limb length, knee and ankle joint width, width and depth of the pelvis). Whole gait analysis will be performed by experienced single clinical biomechanist accordingly to the Davis protocol. Markers will be installed on the patients' limbs on the following points: base of sacral bone, greater trochanter of the femur, lateral femoral condyle, head of the fibula, lateral malleoli, head of the V metatarsal bone).

Participants will walk barefoot for 10 meters quadruple times. Following time-space and kinematic parameters will be assessed:

Time-space parameters Single stance time (T1) [%] Swing time (T2) [%] Double-stance time (T3) [%] Step length (SL) [m] Mean gait velocity (Vm) [m/s] Cadence (C) [number of steps/min]

Kinematic parameters:

Operated knee range of flexion during swing phase [°]

ELIGIBILITY:
Inclusion Criteria:

* agreement to participate in the study
* BMI (kg/m2) less than 40
* ability to walk for 10 meters
* knee flexion more or equal of 90 degrees

Exclusion Criteria:

* unwillingness to participate in the study
* osteoarthritis due to the rheumatological disease
* disorders associated with nerve-muscle signal transmission
* neurological disorders associated with dizziness, nystagmus or other conditions that might influence balance during activity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
Time of swing phase | Time Frame: 1-3 years after surgery
  Change from baseline part of swing phase time during gait, measured in percentage
  Change from baseline part of swing phase time during gait, measured in percentage
Time of stance phase | Time Frame: 1-3 years after surgery
  Change from baseline part of stance phase time during gait, measured in percentage
Time of double-stance phase | Time Frame: 1-3 years after surgery
  Change from baseline part of double-stance phase time during gait, measured in percentage
Stride length | Time Frame: 1-3 years after surgery
  Change from baseline length of stride during gait, measured in meters
Cadence | Time Frame: 1-3 years after surgery
  Change from baseline number of strides per minute of walking
Mean gait velocity | Time Frame: 1-3 years after surgery
  Change from baseline mean values of gait speed, measured in meters per second
Range of maximal hip extension for both limbs during ending part of mid-stance phase | Time Frame: 1-3 years after surgery
  Change from baseline range of maximal hip extension for both limbs during ending part of mid-stance phase, measured in degrees
Range of pelvic drop in frontal plane on the opposite site of the bearing limb | Time Frame: 1-3 years after surgery
  Change from baseline range of pelvic drop in frontal plane on the opposite site of the bearing limb, measured in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz M. Maciąg, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland